CLINICAL TRIAL: NCT04846439
Title: Sequential Infusion of CD19 and BCMA Chimeric Antigen Receptor T Cells to Improve Alloimmune-mediated Platelet Transfusion Refractoriness in Patients With Acute Leukemia in Complete Remission
Brief Title: Sequential Infusion of CD19 and BCMA CAR-T Cells to Improve PTR in Patients With AL
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: The Second People's Hospital of Huai'an (Other); The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Shanghai Unicar-Therapy Bio-medicine Technology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021062
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-04

CONDITIONS: Platelet Transfusion Refractoriness; Acute Leukemia in Remission
Keywords: CAR-T; alloimmune; platelet transfusion refractoriness
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T infusion (Experimental): CD19 and BCMA CAR-T cells were infused into complete remission acute leukemia patients with PTR sequentially, with（1.0-2.0）×10e7/kg respectively. Each patient was followed up for 1 years.
  Interventions: Biological: CAR-T infusion

INTERVENTIONS:
Biological: CAR-T infusion — Sequential infusion of CD19 and BCMA autologous chimeric antigen receptor T cells, the infusion dose was determined according to the body weight of the subject and the effective content of cell preparation.

SUMMARY:
Alloimmune-mediated platelet transfusion refractoriness(PTR) was usually caused by repeated blood transfusions and pregnancy and accounts for about 20-25% of PTR patients. Patients with acute leukemia need repeated platelet infusion in myelosuppression period after chemotherapy, and PTR incidence is more higher.PTR was associated with adverse events,including longer hospital stays,severe hemorrhages and an increased risk of early deaths and may have a negative impact on the success of HSCT. The current management of patients with PTR includes specific transfusion strategies, IVIG, rituximab,thrombopoietin-receptor agonists(TPO-RA) ,bortezomib or splenectomy,have been largely unsatisfactory. As we know, HLA antibodies are mainly secreted by the plasma cells. Researchers want to see if sequential infusion of CD19 and BCMA CAR-T cells can clear the B cells and plasma cells, can help increase platelet levels and reduce bleeding in patients with platelet transfusion refractoriness. To see if sequential infusion can increases platelet levels more after a transfusion. To see if it reduces the chance of bleeding. Adults 16-65 years old who diagnosed with acute leukemia in CR and alloimmune platelet transfusion refractoriness.

DETAILED DESCRIPTION:
The patients will receive infusion of CAR T-cells targeting CD19 and BCMA to confirm the safety and efficacy of CD19 and BCMA CAR T-Cells Sequential infusion in acute leukemia with alloimmune-mediated platelet transfusion refractoriness.

ELIGIBILITY:
Inclusion Criteria:

* Ages 16-65 years inclusive.
* Ability to comprehend the investigational nature of the study and provide informed consent.
* Expected survival time ≥ 3 months (according to investigator's judgement)
* Acute leukemia in complete remission diagnosed with alloimmune-mediated PTR, characterized by all of the following:

Lack of adequate post-transfusion platelet count increment, defined by CCI <7500/μl at 10-60 min, and CCI <5000/μl at 18-24 hrs (in those who had a CCI at 10-60 min greater than or equal to 5000/μl) after at least 2 consecutive transfusions.

Presence of anti-HLA class A and/or B antibody.

* Left ventricular ejection fractions ≥ 0.5 by echocardiography.
* Creatinine < 1.6 mg/dL.
* Aspartate aminotransferase/aspartate aminotransferase < 3x upper limit of normal.
* Total bilirubin <2.0 mg/dL.
* karnofsky performance status ≥ 60.

Exclusion Criteria:

* PTR induced by other reasons(eg:DIC,fever,infection and splenomegaly)
* Uncontrolled active infection.
* Active hepatitis B or hepatitis C infection
* Patients with HIV or syphilis infection
* Patients are pregnant or lactating
* Patients has a history of allo-HSCT
* Alloimmune-mediated PTR responsive to treatment with plasma exchange
* Alloimmune-mediated PTR responsive to treatment with rituximab or IVIG
* Grade III/IV cardiovascular disability according to the New York Heart Association Classification
* Patients with other contraindications considered unsuitable for participation in this study (according to investigator's judgement)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects With Sustained Platelet Transfusion Responsiveness | 12 months
  To evaluate the safety and efficacy of sequential infusion of CD19 and BCMA CAR-T cells to improve PTR, estimate by platelet increment, defined as Corrected Count Increment (CCI) >7500/μL at 10-60 min together with CCI>5000/μL at 18-24 hrs post platelet transfusion in patients with platelet transfusion refractoriness.
Adverse events after sequential infusion of CAR-T | 12 months
  Adverse events are evaluated with CTCAE V5.0.

SECONDARY OUTCOMES:
B lymphocytes/plasma cell clearance | 12 months
  To investigate the possible mechanisms of sequential infusion in alloimmune-mediated PTR
Amplification,distribution and persistence of CAR T-cells in vivo | 12 months
  To evaluate the persistence of CAR-T cells in vivo
Alloimmune antibodies(include HLA and HPA) in PB after sequential transfusion | 12 months
  To evaluate the clearance of alloimmune antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Haiping Dai, Ph.D, Principal Investigator — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China